CLINICAL TRIAL: NCT07213726
Title: Quantification of Peripheral Hematopoietic Progenitor Cell Circulation Following Repeated Acute, Vascular Restriction Resistance Exercise Using the Delfi Tourniquet System
Brief Title: Quantification of Progenitor Cell Circulation Following Vascular Resistance Exercise Using Delfi Tourniquet System
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Andrews Research & Education Foundation (Other)
Collaborators: Florida (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: Extended Delfi
Record Dates: First submitted 2022-10-28; First posted 2025-10-09 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-12

CONDITIONS: Blood Flow Restriction (BFR) Training Effects

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Healthy (Experimental): This group consists of all participants in this study. Subjects must be healthy, and gender is not a factor for enrollment.
  Interventions: Device: Delfi Personalized Tourniquet System

INTERVENTIONS:
Device: Delfi Personalized Tourniquet System — Bilateral proximal thigh bands that will be applied and inflated to a pressure of 80% of occlusive pressure as determined by the automated tourniquet before exercise. A standard exercise session would not include any blood occlusion.

SUMMARY:
The purpose of this observational study is to examine how slowing down blood flow to the legs- a practice called blood flow restriction (BFR)- during exercise by applying compression to the legs affects the way stem cells are released into the blood stream. This will be determined by drawing 6 cubic centimeters (ccs) of blood immediately post-exercise after the Delfi Personalized Tourniquet System (PTS) has been removed. 6 ccs of blood will also be taken prior to exercise and at the 20-, 40-, and 60-minute marks after exercise. The main question of this study is:

• Will the levels of stem cells extracted before and after exercise be the same if blood flow is restricted during exercise?

In this study, participants will undergo the following:

* 6 ccs of blood extracted from the forearm prior to exercise to establish a baseline
* 3 exercises- seated leg extension, semi-reclined leg press, and seated hamstring curl- consisting of 4 sets of 30-15-15-15 repetitions per exercise; resistance will be set to 30% of one-rep maximum (1-RM)
* Additional 6 cc blood draws will be performed immediately post-exercise and after 20, 40, and 60 minutes have elapsed

DETAILED DESCRIPTION:
The proposed study is a prospective, quasi-experiment, dual-center (exercise facility and laboratory) study involving 15 healthy, male and female volunteers. A potential subject must clear the screening, consent to the procedures of this study, and complete the medical interview before proceeding with the familiarization session. The familiarization process will include an introduction to the Delfi BFR Tourniquet System (Delfi Medical Innovations Inc., Vancouver, BC) and the exercises (seated leg extension, semi-reclined leg press, seated hamstring curl) that the subject will complete. The weight each subject will use for each exercise will be determined during this time. All familiarization procedures must be completed prior to the scheduling and execution of the first of twelve experimental testing sessions.

The experimental testing sessions will occur twice a week for six weeks (12 sessions) and will involve the BFR training utilizing the Delfi BFR Tourniquet System, as further described in the Experimental Testing Session section of the treatment plan (6.2). At the beginning of the first, the sixth, and the twelfth testing sessions there will be a blood draw requiring 6 cc of blood to be taken prior to exercise. Post-exercise, at each testing session, additional 6cc blood draws will be conducted immediately post exercise (time point 0), as well as 20- , 40- , and 60 minutes after the conclusion of the workout. Following every testing session workout, finger-prick blood samples for lactate testing will be taken. These blood samples are to be taken at Time point 0- (T 0), 10-, 20-, 30-, 40-, 50-, and 60-minutes following exercise. Once the twelfth experimental testing session has been completed, the subjects will have one final session that is to take place no more than five days following the twelfth testing session. This final session will include one final blood draw of 6 cc. Throughout the duration of the study, the blood drawn will be used for obtaining a complete blood count (CBC) and for cellular analysis to quantify peripheral hematopoietic progenitor cell concentration. The blood samples collected from subject's fingers throughout the study will be used for analysis using a portable lactate analyzer. Lactate analysis will allow researchers insight into each subject's exertion level reflected by the amount of lactate found within the samples collected.

ELIGIBILITY:
Inclusion Criteria

1. Volunteer population of healthy males and females aged 18-45.
2. Subjects consent to attending a total of 14 visits over a time span of seven to nine weeks. The breakdown of the 14 visits is as follows: 1 familiarization session, 12 experimental testing sessions, 1 final session.

Exclusion Criteria

Volunteers who have medical history involving one or more of the following medical conditions:

1. Diabetes
2. Uncontrolled hypertension
3. Autoimmune disorders
4. Blood disorders
5. Ongoing infectious disease
6. Cancer
7. Any disorder requiring immunosuppression treatment
8. Steroid usage
9. Significant cardiovascular, pulmonary, hepatic, or renal disease.
10. Volunteers where 20 minutes of intense exercise is contra-indicated will also be excluded from the study.
11. Positive pregnancy test

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Estimated)
Dates: Start 2022-08-16 (Actual); Primary Completion 2023-11-20 (Actual); Study Completion 2026-11-20 (Estimated)

PRIMARY OUTCOMES:
Concentration of Blood Lactate | 1 week after enrollment
  Allows researchers insight into each subject's exertion level reflected by the amount of lactate found within the samples collected.
Concentration of Blood Lactate | 2 weeks after enrollment
  Allows researchers insight into each subject's exertion level reflected by the amount of lactate found within the samples collected.
Concentration of Blood Lactate | 3 weeks after enrollment
  Allows researchers insight into each subject's exertion level reflected by the amount of lactate found within the samples collected.
Concentration of Blood Lactate | 4 weeks after enrollment
  Allows researchers insight into each subject's exertion level reflected by the amount of lactate found within the samples collected.
Concentration of Blood Lactate | 5 weeks after enrollment
  Allows researchers insight into each subject's exertion level reflected by the amount of lactate found within the samples collected.
Concentration of Blood Lactate | 6 weeks after enrollment
  Allows researchers insight into each subject's exertion level reflected by the amount of lactate found within the samples collected.
Prevalence of Hematopoietic Stem Cells | 1 week after enrollment
  Technique completed using special machine that utilizes lasers to separate and quantify various content of cell samples; used in this study to determine complete blood cell count (CBC) and peripheral hematopoietic progenitor cell concentration
Prevalence of Hematopoietic Stem Cells | 2 weeks after enrollment
  Technique completed using special machine that utilizes lasers to separate and quantify various content of cell samples; used in this study to determine complete blood cell count (CBC) and peripheral hematopoietic progenitor cell concentration
Prevalence of Hematopoietic Stem Cells | 3 weeks after enrollment
  Technique completed using special machine that utilizes lasers to separate and quantify various content of cell samples; used in this study to determine complete blood cell count (CBC) and peripheral hematopoietic progenitor cell concentration
Prevalence of Hematopoietic Stem Cells | 4 weeks after enrollment
  Technique completed using special machine that utilizes lasers to separate and quantify various content of cell samples; used in this study to determine complete blood cell count (CBC) and peripheral hematopoietic progenitor cell concentration
Prevalence of Hematopoietic Stem Cells | 5 weeks after enrollment
  Technique completed using special machine that utilizes lasers to separate and quantify various content of cell samples; used in this study to determine complete blood cell count (CBC) and peripheral hematopoietic progenitor cell concentration
Prevalence of Hematopoietic Stem Cells | 6 weeks after enrollment
  Technique completed using special machine that utilizes lasers to separate and quantify various content of cell samples; used in this study to determine complete blood cell count (CBC) and peripheral hematopoietic progenitor cell concentration

CONTACTS AND LOCATIONS:
Overall Officials: Tyler Opitz, DPT, SCS, CSCS, Principal Investigator — Physical Therapist
Locations (1):
- Andrews Institute for Orthopaedics & Sports Medicine, Gulf Breeze, Florida, United States

REFERENCES:
- [Background] Weissman IL, Shizuru JA. The origins of the identification and isolation of hematopoietic stem cells, and their capability to induce donor-specific transplantation tolerance and treat autoimmune diseases. Blood. 2008 Nov 1;112(9):3543-53. doi: 10.1182/blood-2008-08-078220. PMID 18948588
- [Background] Zakrzewski JL, van den Brink MR, Hubbell JA. Overcoming immunological barriers in regenerative medicine. Nat Biotechnol. 2014 Aug;32(8):786-94. doi: 10.1038/nbt.2960. PMID 25093888
- [Background] Caplan AI. Mesenchymal stem cells. J Orthop Res. 1991 Sep;9(5):641-50. doi: 10.1002/jor.1100090504. PMID 1870029
- [Background] Marycz K, Mierzejewska K, Smieszek A, Suszynska E, Malicka I, Kucia M, Ratajczak MZ. Endurance Exercise Mobilizes Developmentally Early Stem Cells into Peripheral Blood and Increases Their Number in Bone Marrow: Implications for Tissue Regeneration. Stem Cells Int. 2016;2016:5756901. doi: 10.1155/2016/5756901. Epub 2015 Nov 9. PMID 26664409
- [Background] Agha NH, Baker FL, Kunz HE, Graff R, Azadan R, Dolan C, Laughlin MS, Hosing C, Markofski MM, Bond RA, Bollard CM, Simpson RJ. Vigorous exercise mobilizes CD34+ hematopoietic stem cells to peripheral blood via the beta2-adrenergic receptor. Brain Behav Immun. 2018 Feb;68:66-75. doi: 10.1016/j.bbi.2017.10.001. Epub 2017 Oct 7. PMID 29017969
- [Background] Callanan MC, Plummer HA, Chapman GL, Opitz TJ, Rendos NK, Anz AW. Blood Flow Restriction Training Using the Delfi System Is Associated With a Cellular Systemic Response. Arthrosc Sports Med Rehabil. 2020 Dec 27;3(1):e189-e198. doi: 10.1016/j.asmr.2020.09.009. eCollection 2021 Feb. PMID 33615264
- [Background] Hwang NS, Zhang C, Hwang YS, Varghese S. Mesenchymal stem cell differentiation and roles in regenerative medicine. Wiley Interdiscip Rev Syst Biol Med. 2009 Jul-Aug;1(1):97-106. doi: 10.1002/wsbm.26. PMID 20835984
- [Background] Docheva D, Popov C, Mutschler W, Schieker M. Human mesenchymal stem cells in contact with their environment: surface characteristics and the integrin system. J Cell Mol Med. 2007 Jan-Feb;11(1):21-38. doi: 10.1111/j.1582-4934.2007.00001.x. PMID 17367499
- [Background] Rochefort GY, Delorme B, Lopez A, Herault O, Bonnet P, Charbord P, Eder V, Domenech J. Multipotential mesenchymal stem cells are mobilized into peripheral blood by hypoxia. Stem Cells. 2006 Oct;24(10):2202-8. doi: 10.1634/stemcells.2006-0164. Epub 2006 Jun 15. PMID 16778152
- [Background] Hylden C, Burns T, Stinner D, Owens J. Blood flow restriction rehabilitation for extremity weakness: a case series. J Spec Oper Med. 2015 Spring;15(1):50-6. PMID 25770798
- [Background] Takarada Y, Takazawa H, Ishii N. Applications of vascular occlusion diminish disuse atrophy of knee extensor muscles. Med Sci Sports Exerc. 2000 Dec;32(12):2035-9. doi: 10.1097/00005768-200012000-00011. PMID 11128848
- [Background] Vechin FC, Libardi CA, Conceicao MS, Damas FR, Lixandrao ME, Berton RP, Tricoli VA, Roschel HA, Cavaglieri CR, Chacon-Mikahil MP, Ugrinowitsch C. Comparisons between low-intensity resistance training with blood flow restriction and high-intensity resistance training on quadriceps muscle mass and strength in elderly. J Strength Cond Res. 2015 Apr;29(4):1071-6. doi: 10.1519/JSC.0000000000000703. PMID 25264670
- [Background] Takarada Y, Takazawa H, Sato Y, Takebayashi S, Tanaka Y, Ishii N. Effects of resistance exercise combined with moderate vascular occlusion on muscular function in humans. J Appl Physiol (1985). 2000 Jun;88(6):2097-106. doi: 10.1152/jappl.2000.88.6.2097. PMID 10846023
- [Background] Feriche B, Garcia-Ramos A, Morales-Artacho AJ, Padial P. Resistance Training Using Different Hypoxic Training Strategies: a Basis for Hypertrophy and Muscle Power Development. Sports Med Open. 2017 Dec;3(1):12. doi: 10.1186/s40798-017-0078-z. Epub 2017 Mar 17. PMID 28315193
- [Background] Kaijser L, Sundberg CJ, Eiken O, Nygren A, Esbjornsson M, Sylven C, Jansson E. Muscle oxidative capacity and work performance after training under local leg ischemia. J Appl Physiol (1985). 1990 Aug;69(2):785-7. doi: 10.1152/jappl.1990.69.2.785. PMID 2146245
- [Background] Farup J, de Paoli F, Bjerg K, Riis S, Ringgard S, Vissing K. Blood flow restricted and traditional resistance training performed to fatigue produce equal muscle hypertrophy. Scand J Med Sci Sports. 2015 Dec;25(6):754-63. doi: 10.1111/sms.12396. Epub 2015 Jan 21. PMID 25603897
- [Background] Ellefsen S, Hammarstrom D, Strand TA, Zacharoff E, Whist JE, Rauk I, Nygaard H, Vegge G, Hanestadhaugen M, Wernbom M, Cumming KT, Ronning R, Raastad T, Ronnestad BR. Blood flow-restricted strength training displays high functional and biological efficacy in women: a within-subject comparison with high-load strength training. Am J Physiol Regul Integr Comp Physiol. 2015 Oct;309(7):R767-79. doi: 10.1152/ajpregu.00497.2014. Epub 2015 Jul 22. PMID 26202071
- [Background] de Freitas MC, Gerosa-Neto J, Zanchi NE, Lira FS, Rossi FE. Role of metabolic stress for enhancing muscle adaptations: Practical applications. World J Methodol. 2017 Jun 26;7(2):46-54. doi: 10.5662/wjm.v7.i2.46. eCollection 2017 Jun 26. PMID 28706859
- [Background] Vanwye WR, Weatherholt AM, Mikesky AE. Blood Flow Restriction Training: Implementation into Clinical Practice. Int J Exerc Sci. 2017 Sep 1;10(5):649-654. doi: 10.70252/LYGQ7085. eCollection 2017. PMID 28966705
- [Background] Loenneke JP, Fahs CA, Rossow LM, Abe T, Bemben MG. The anabolic benefits of venous blood flow restriction training may be induced by muscle cell swelling. Med Hypotheses. 2012 Jan;78(1):151-4. doi: 10.1016/j.mehy.2011.10.014. Epub 2011 Nov 1. PMID 22051111
- [Background] Wilson JM, Lowery RP, Joy JM, Loenneke JP, Naimo MA. Practical blood flow restriction training increases acute determinants of hypertrophy without increasing indices of muscle damage. J Strength Cond Res. 2013 Nov;27(11):3068-75. doi: 10.1519/JSC.0b013e31828a1ffa. PMID 23446173
- [Background] Loenneke JP, Abe T, Wilson JM, Thiebaud RS, Fahs CA, Rossow LM, Bemben MG. Blood flow restriction: an evidence based progressive model (Review). Acta Physiol Hung. 2012 Sep;99(3):235-50. doi: 10.1556/APhysiol.99.2012.3.1. PMID 22982712
- [Background] Reeves GV, Kraemer RR, Hollander DB, Clavier J, Thomas C, Francois M, Castracane VD. Comparison of hormone responses following light resistance exercise with partial vascular occlusion and moderately difficult resistance exercise without occlusion. J Appl Physiol (1985). 2006 Dec;101(6):1616-22. doi: 10.1152/japplphysiol.00440.2006. Epub 2006 Aug 10. PMID 16902061
- [Background] Inagaki Y, Madarame H, Neya M, Ishii N. Increase in serum growth hormone induced by electrical stimulation of muscle combined with blood flow restriction. Eur J Appl Physiol. 2011 Nov;111(11):2715-21. doi: 10.1007/s00421-011-1899-y. Epub 2011 Mar 12. PMID 21399959
- [Background] Schoenfeld BJ. Potential mechanisms for a role of metabolic stress in hypertrophic adaptations to resistance training. Sports Med. 2013 Mar;43(3):179-94. doi: 10.1007/s40279-013-0017-1. PMID 23338987
- [Background] Pearson SJ, Hussain SR. A review on the mechanisms of blood-flow restriction resistance training-induced muscle hypertrophy. Sports Med. 2015 Feb;45(2):187-200. doi: 10.1007/s40279-014-0264-9. PMID 25249278
- [Background] Manini TM, Yarrow JF, Buford TW, Clark BC, Conover CF, Borst SE. Growth hormone responses to acute resistance exercise with vascular restriction in young and old men. Growth Horm IGF Res. 2012 Oct;22(5):167-72. doi: 10.1016/j.ghir.2012.05.002. Epub 2012 Jun 23. PMID 22727808
- [Background] Takano H, Morita T, Iida H, Asada K, Kato M, Uno K, Hirose K, Matsumoto A, Takenaka K, Hirata Y, Eto F, Nagai R, Sato Y, Nakajima T. Hemodynamic and hormonal responses to a short-term low-intensity resistance exercise with the reduction of muscle blood flow. Eur J Appl Physiol. 2005 Sep;95(1):65-73. doi: 10.1007/s00421-005-1389-1. Epub 2005 Jun 15. PMID 15959798
- [Background] Takarada Y, Nakamura Y, Aruga S, Onda T, Miyazaki S, Ishii N. Rapid increase in plasma growth hormone after low-intensity resistance exercise with vascular occlusion. J Appl Physiol (1985). 2000 Jan;88(1):61-5. doi: 10.1152/jappl.2000.88.1.61. PMID 10642363
- [Background] Ganesan G, Cotter JA, Reuland W, Cerussi AE, Tromberg BJ, Galassetti P. Effect of blood flow restriction on tissue oxygenation during knee extension. Med Sci Sports Exerc. 2015 Jan;47(1):185-93. doi: 10.1249/MSS.0000000000000393. PMID 24870580
- [Background] Scott BR, Slattery KM, Sculley DV, Dascombe BJ. Hypoxia and resistance exercise: a comparison of localized and systemic methods. Sports Med. 2014 Aug;44(8):1037-54. doi: 10.1007/s40279-014-0177-7. PMID 24715613
- [Background] Narici MV, Kayser B. Hypertrophic response of human skeletal muscle to strength training in hypoxia and normoxia. Eur J Appl Physiol Occup Physiol. 1995;70(3):213-9. doi: 10.1007/BF00238566. PMID 7607195

DOCUMENTS (2):
  • Study Protocol (2022-11-01): https://cdn.clinicaltrials.gov/large-docs/26/NCT07213726/Prot_000.pdf
  • Informed Consent Form (2022-08-08): https://cdn.clinicaltrials.gov/large-docs/26/NCT07213726/ICF_001.pdf